CLINICAL TRIAL: NCT00002406
Title: A Multicenter, Open-Label, Randomized, 24-Week Study to Compare the Safety and Activity of Indinavir Sulphate, 800 Mg q 8h Versus 1,200 Mg q 12h in HIV-Infected Individuals Having Plasma Viral RNA Less Than 400 Copies/Ml, on Concomitant Therapy With 2 Nucleoside Analogue Reverse Transcriptase Inhibitors (NRTI)
Brief Title: A Comparison of Two Dose Levels of Indinavir Combined With Two Nucleoside Analogue Reverse Transcriptase Inhibitors (NRTIs) in HIV-Infected Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: None | Purpose: Treatment
Other Study IDs: 246P; MK-0639
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-06

CONDITIONS: HIV Infections
Keywords: HIV-1; Dose-Response Relationship, Drug; HIV Protease Inhibitors; Indinavir; RNA, Viral; Reverse Transcriptase Inhibitors
MeSH Terms: conditions — HIV Infections | interventions — Indinavir

INTERVENTIONS:
Drug: Indinavir sulfate

SUMMARY:
The purpose of this study is to determine if two dose levels of indinavir combined with two nucleoside analogue reverse transcriptase inhibitors (NRTIs) have the same effect on plasma viral load (level of HIV in the blood).

DETAILED DESCRIPTION:
In this open-label study 350 seropositive HIV-1 men and women are first stratified according to baseline plasma viral RNA (less than 400 copies/mL vs negative plasma viral RNA result) then randomized into one of two arms:

Arm 1: Indinavir (800 mg, q8h) plus two pre-existing NRTIs. Arm 2: Indinavir (1,200 mg, q12h) plus two pre-existing NRTIs. Plasma viral RNA will be measured every 4 weeks for the duration of the 24-week study.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* Documented HIV-1 seropositive status.
* CD4 count greater than 100 cells/mm3.
* Parental consent for patients under 18.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350

CONTACTS AND LOCATIONS:
Locations (29):
- United States (29):
  - 1917 Research Clinic, Birmingham, Alabama
  - Kaiser Permanente / Infectious Disease, Los Angeles, California
  - Tower ID Med Associates, Los Angeles, California
  - Ctr for AIDS Research / Education and Service (CARES), Sacramento, California
  - San Francisco Gen Hosp / UCSF AIDS Program, San Francisco, California
  - HIV Clinical Research, Fort Lauderdale, Florida
  - Univ of Miami School of Medicine, Miami, Florida
  - AIDS Research Consortium of Atlanta, Atlanta, Georgia
  - Ponce de Leon Ctr, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Rush Presbyterian St Lukes Med Ctr, Chicago, Illinois
  - Natl Naval Med Ctr / Special Immunology Clinic, Bethesda, Maryland
  - Brigham and Women's Hosp, Boston, Massachusetts
  - Boston Med Ctr / Clinical Research Office, Boston, Massachusetts
  - Univ Health Ctr 7D, Detroit, Michigan
  - Kansas City Free Health Clinic, Kansas City, Missouri
  - Education & Research Building, Camden, New Jersey
  - Garden State Infectious Diseases / E I P Kennedy Health Sys, Voorhees Township, New Jersey
  - Albany Med College / Div of HIV Medicine, Albany, New York
  - SUNY / Health Science Ctr at Brooklyn, Brooklyn, New York
  - New York Hosp of Queens / AIDS Ctr, Flushing, New York
  - CRIA, New York, New York
  - St Vincents Hosp and Med Ctr / Div of HIV Med, New York, New York
  - Anderson Clinical Research, New York, New York
  - Akron City Hospital, Akron, Ohio
  - Thomas Jefferson Univ, Philadelphia, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Houston Clinical Research Network / Southhampton Med Group, Houston, Texas
  - Univ of Utah School Of Medicine / Div of Infec Disease, Salt Lake City, Utah